CLINICAL TRIAL: NCT07318558
Title: A Phase 3, Randomized, Open-label, Multicenter Study of Sacituzumab Tirumotecan (Sac-TMT, MK-2870) Maintenance Treatment With or Without Bevacizumab Versus Standard of Care in Participants With Newly Diagnosed Advanced HRD-Negative Ovarian Cancer Following First-line Platinum-based Chemotherapy (TroFuse-021/ENGOTov85/GOG-3102)
Brief Title: A Clinical Trial of Sacituzumab Tirumotecan in People With Ovarian Cancer (MK-2870-021)
Acronym: TroFuse-021
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2870-021; MK-2870-021 (Other: MSD); GOG-3102 (Other: Gynecologic Oncology Group); ENGOT-ov85 (Other: European Network for Gynaecological Oncological Trial groups)
Record Dates: First submitted 2026-01-02; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Neoplasms; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sac-TMT +/- Bevacizumab (Experimental): Participants will receive sac-TMT on days 1, 15, and 29 (q2W) of every 6-week cycle, until disease progression, prohibitive toxicity, or other protocol-defined reason for discontinuation. Participants receive optional bevacizumab at investigator's discretion on Days 1 and 22 (q3w) of every 6-week cycle, for up to 22 courses.
  Interventions: Drug: Sacituzumab tirumotecan; Drug: Bevacizumab; Drug: Rescue Medications
- Standard of Care (Active Comparator): Participants will either receive bevacizumab q3w of every 6-week cycle for up to 22 courses until disease progression, prohibitive toxicity, or other protocol-defined reason for discontinuation of study intervention, or will be observed only and actively followed if not receiving bevacizumab.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Sacituzumab tirumotecan — Administered via intravenous (IV) infusion at a dose of 4mg/kg
  Other Names: sac-TMT; MK-2870; SKB264
  Arms: Sac-TMT +/- Bevacizumab
Drug: Bevacizumab — Administered via IV infusion at a dose of 15mg/kg
  Other Names: Avastin; Altuzan; MVASI
Drug: Rescue Medications — Participants receive the following rescue medications prior to sac-TMT infusion, per approved product label: histamine-1 receptor antagonist, histamine-2 receptor antagonist, acetaminophen or equivalent, and dexamethasone or equivalent. Participants are also recommended to receive prophylactic steroid mouthwash (dexamethasone or equivalent).
  Arms: Sac-TMT +/- Bevacizumab

SUMMARY:
Researchers are looking for new ways to treat ovarian cancer (OC). Current treatment for OC may start with surgery to remove as much of the cancer as possible. After surgery, people may receive chemotherapy. After chemotherapy, standard care options may include:

* Maintenance treatment, which is used after another therapy to keep the cancer from growing, spreading, or coming back. Bevacizumab is a targeted therapy used as standard maintenance treatment. Targeted therapy works to control how specific types of cancer cells grow and spread.
* Observation, which is watching to see if cancer grows or worsens

The study medicine, sacituzumab tirumotecan (also called sac-TMT), is a targeted therapy. The goal of this study is to learn if people who receive sac-TMT maintenance treatment with or without bevacizumab live longer without the cancer getting worse than people who receive standard care.

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Has histologically confirmed epithelial ovarian, primary peritoneal, or fallopian tube cancer.
* Has completed primary debulking surgery or interval debulking surgery.
* Has completed first-line (1L) platinum-based chemotherapy, with a response of stable disease, partial response, or complete response per protocol.
* Has provided tumor tissue that is not previously irradiated.
* If human immunodeficiency virus (HIV) infected, has well-controlled HIV on antiretroviral therapy.
* Has undetectable hepatitis B virus (HBV) viral load and received HBV antiviral therapy if hepatitis B surface antigen (HBsAg)-positive.
* Has undetectable hepatitis C virus (HCV) viral load if has a history of HCV infection.

The main exclusion criteria include but are not limited to the following:

* Has nonepithelial cancers, borderline tumors mucinous, seromucinous that is predominantly mucinous, malignant Brenner's tumor, and undifferentiated carcinoma.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has a history of severe eye disease.
* Has active inflammatory bowel disease requiring immunosuppressive medication or a previous history of inflammatory bowel disease.
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease (ILD), which required steroids, or has current pneumonitis/ILD.
* Received prior systemic anticancer therapy, with the exception of the first-line platinum-based chemotherapy required by the inclusion criteria.
* Had a live or live-attenuated vaccine within 30 days of randomization.
* Has a known additional malignancy that is progressing or required active treatment within the past 3 years.
* Has active infection requiring systemic therapy.
* Has concurrent and active HBV and HCV infections.
* Has HIV infection and a history of Kaposi's sarcoma and/or multicentric Castleman's disease.
* Has not recovered from major surgery or has ongoing surgical complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 900 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2033-02-25 (Estimated); Study Completion 2033-05-20 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 49 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 by blinded independent central review (BICR) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 78 months
  OS is defined as the time from randomization to death due to any cause.
Progression-Free Survival 2 (PFS2) | Up to approximately 78 months
  PFS2 as assessed by investigator is defined as the time from randomization to the documented subsequent objective disease progression after initiation of new anticancer therapy or death due to any cause, whichever occurs first.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 78 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 78 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Change From Baseline in Global Health Status/Quality of Life (GHS/QoL) Combined Score (Items 29 and 30) Using the European Organisation for Research and Treatment of Cancer QoL Questionnaire-Core 30 (EORTC QLQ-C30) | Baseline, and at designated time points up to approximately 78 months
  EORTC QLQ-C30 is a questionnaire to assess the overall quality of life (QoL) of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7- point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.
Change From Baseline in Physical Functioning Combined Score (Items 1 to 5) Using EORTC QLQ-C30 | Baseline, and at designated time points up to approximately 78 months
  EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1 = Not at All to 4 = Very Much). The combined score is computed by averaging the raw scores of the 5 questions and then applying a linear transformation to standardize the average score, so that the combined score ranges from 0 to 100. A higher score indicates a better outcome. The change from baseline in the EORTC QLQ-C30 physical functioning combined score will be presented.
Change From Baseline in Role Functioning Combined Score (Items 6 and 7) Using EORTC QLQ-C30 | Baseline, and at designated time points up to approximately 78 months
  EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 2 questions about their role functioning are scored on a 4-point scale (1 = Not at All to 4 = Very Much). The combined score is computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined score ranges from 0 to 100. A higher score indicates a better outcome. The change from baseline in the EORTC QLQ-C30 role functioning combined score will be presented.
Change From Baseline in Abdominal/Gastrointestinal (GI) Symptoms Combined Score Using the EORTC QLQ-Ovarian Cancer Module 28 (OV28) | Baseline, and at designated time points up to approximately 78 months
  EORTC QLQ-OV28 is an OC-specific module to supplement the EORTC QLQ-C30. Participant responses to the 6 abdominal/GI symptoms scale questions are scored on a 4-point scale (1=not at all, 4=very much). The combined score is computed by averaging the raw scores of the 6 items and then applying a linear transformation to standardize the average score, so that the combined score ranges from 0 to 100. The change from baseline in abdominal and gastrointestinal symptoms (EORTC QLQ-OC28 Items 31-36) score will be presented. A lower score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/